CLINICAL TRIAL: NCT06677372
Title: Comparative Analysis of Core Body Temperature Measurement During Endoscopy: Esophageal Temperature Probe Versus Skin Temperature Sensors
Brief Title: Comparative Analysis of Core Body Temperature Measurement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jong Yu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2311-164-1488
Record Dates: First submitted 2024-11-02; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2023-12

CONDITIONS: Temperature Change, Body
Keywords: Esophageal temperature; 3M Spot On; Zero heat flux temperature
MeSH Terms: conditions — Body Temperature Changes | interventions — Body Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Diagnostic Test: Body temperature measurement

INTERVENTIONS:
Diagnostic Test: Body temperature measurement — Comparative analysis of temperature between esophageal temperature and skin temperature

SUMMARY:
Comparison and evaluation of the correlation, accuracy, and precision between a skin-attached temperature sensor and the standard method of deep body temperature measurement, the esophageal thermometer, by measuring and assessing both temperature measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 years and above, but under 70 years

Exclusion Criteria:

* Cases where there were serious side effects during a previous examination performed under sedation or anesthesia
* Currently undergoing treatment for a diagnosed disease
* Diagnosed with esophageal varices or having a history of esophagitis
* Having undergone esophageal and gastric resection surgery

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Body temperature | From enrollment to the end of the treatment at 1month
  Esophageal Temperature Probe versus Skin Temperature Sensors

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No